CLINICAL TRIAL: NCT05617482
Title: Comparison Between Ultrasound-guided Ilioinguinal, Iliohypogastric Nerve Blocks, TAP Block and Quadratus Lumborum Block in Patients Scheduled for Lower Segment Ceserian Sections. A Randomized Controlled Trial
Brief Title: Comparison Between Ultrasound-guided Ilioinguinal, Iliohypogastric Nerve Blocks, TAP Block and Quadratus Lumborum Block in Patients Scheduled for Lower Segment Ceserian Sections.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Mogahed, Associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 35633/8/22
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All patients will be informed about the three tyoes of nerve blocks; the ultrasound guided ilioinguinal, iliohypogastric nerve blocks, TAP block and quadratus lumborum block. and will sign that they agree to have any one of them according to randomization.
  Also the outcome assessor will be unaware about the type of nerve block given to the patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasound guided ilioinguinal, iliohypogastric TAP block (Active Comparator): In ilioinguinal-iliohypogastric block group, the probe will be placed medial to the lateral one-third of the line joining the umbilicus and the anterior superior iliac spine (ASIS). The anterior superior iliac crest, iliacus muscle, internal oblique, transverses abdominis, and the ILIH nerves between them will be identified. After appreciating the sonoanatomy, the ILIH nerve will be approached with the 23-gauge Quincke spinal needle through in-plane technique and 10 ml of 0.25% bupivacaine will be injected all around and the drug spread will be appreciated.
  Interventions: Other: General anesthesia; Other: Ilioinguinal, iliohypogastric nerve blocks
- Ultrasound guided transversus abdominis plane block (Active Comparator): The transducer will be placed at between the lower rib margin and the iliac crest, the 23-gauge Quincke spinal needle needle passed through the external oblique and internal oblique muscle till reaching the transversus abdominis sheet. 20 ml of 0.25% bupivacaine will be injected
  Interventions: Other: General anesthesia; Other: TAP block
- Ultrasound guidedQuadratus lumborum block (Active Comparator): The transducer will be placed at the level of the anterosuperior iliac spine and will move cranially until the 3 abdominal wall muscles will be clearly identified. The external oblique muscle will be followed posterolaterally until its posterior border was visualized (hook sign), leaving underneath the internal oblique muscle, like a roof over the quadratus lumborum muscle. The probe will be tilted down to identify a bright hyperechoic line that corresponded with the middle layer of he thoracolumbar fascia. The needle (21 gauge) will be inserted in plane from anterolateral to posteromedial. The optimal point of injection for the QL block will be determined over the lumbar interfacial triangle using hydrodissection.
  Interventions: Other: General anesthesia; Other: Quadratus lumborum block

INTERVENTIONS:
Other: General anesthesia — All patients undergoing ceaserian section under general anesthesia
Other: Ilioinguinal, iliohypogastric nerve blocks — In ilioinguinal-iliohypogastric block group, the probe will be placed medial to the lateral one-third of the line joining the umbilicus and the anterior superior iliac spine (ASIS). The anterior superior iliac crest, iliacus muscle, internal oblique, transverses abdominis, and the ILIH nerves between them will be identified. After appreciating the sonoanatomy, the ILIH nerve will be approached with the 23-gauge Quincke spinal needle through in-plane technique and 10 ml of 0.25% bupivacaine will be injected all around and the drug spread will be appreciated.
  Arms: Ultrasound guided ilioinguinal, iliohypogastric TAP block
Other: TAP block — In TAP block group, the probe will be placed perpendicular to the mid-axillary line between the iliac crest and the subcostal margin and the three abdominal muscle layers will be identified, and the transverses abdominis plane will be located between the internal oblique and the transverse abdominis muscle. The TAP will be approached through in-plane technique using a 23-gauge Quincke spinal needle attached to a 20 ml syringe of 0.25% bupivacaine will be injected and the drug spread in the plane will be observed.
  Arms: Ultrasound guided transversus abdominis plane block
Other: Quadratus lumborum block — For the QLB, the transducer will be placed at the level of the anterosuperior iliac spine and will move cranially until the 3 abdominal wall muscles will be clearly identified. The external oblique muscle will be followed posterolaterally until its posterior border was visualized (hook sign), leaving underneath the internal oblique muscle, like a roof over the quadratus lumborum muscle. The probe will be tilted down to identify a bright hyperechoic line that corresponded with the middle layer of he thoracolumbar fascia. The needle (21 gauge) will be inserted in plane from anterolateral to posteromedial. The optimal point of injection for the QL block will be determined over the lumbar interfacial triangle using hydrodissection.
  Arms: Ultrasound guidedQuadratus lumborum block

SUMMARY:
To compare between Ultrasound guided ilioinguinal, iliohypogastric nerve blocks, TAP block and Quadratus lumborum block in patients scheduled for lower segment ceserian sections.

DETAILED DESCRIPTION:
One hundred and fifty patients belonging to the American Society of Anesthesiologists physical status 1 and 2, aged between 18 and 45 years and will be scheduled for emergency or elective lower segment cesarean section (LSCS) under general anesthesia will be selected between (December 2022 to March 2023, written informed consent will be obtained from all participants.

Inclusion criteria: ASA 1& 2, Age between 18 and 45 years , scheduled for emergency or elective CS under spinal anesthesia; While exclusion criteria:pregnant women who will refuse to participate, known allergy to local anesthetic, infection at the block site.

Patients who will not willing to give consent, known allergy to local anesthetic or infection at the block site will be excluded from the study.

All patients will receive standard premedication according to institute protocol with ranitidine and metoclopramide intravenously immediately before shifting the patient into the operating room for emergency LSCS or 2 h before by oral route in case of elective LSCS. Inside the operating room under all aseptic precautions, spinal anesthesia will be administered using 1.8 ml of 0.5% of heavy bupivacaine without any adjuvant in L3-L4 space using Quincke's needle by the attending anesthesiologist. The case will be managed by the same person without any narcotics intraoperatively. At the end of the procedure just before the skin closure, 1 g of injection paracetamol will be administered intravenously over a period of 20 min as a part of multimodal analgesia. At the end of the surgery, patients will be randomized into ILIH (50 patients) , TAP block group (35 patients) or quadratus lumborum group (50 patients) by choosing a closed envelope, which will contain a standard data collection sheet and an allocation card. All the blocks were performed by the principle investigator under aseptic precautions and ultrasound guidance using high frequency linear probe resonating at 12 MHz in the multi-beam mode. In TAP block group, the probe will be placed perpendicular to the mid-axillary line between the iliac crest and the subcostal margin and the three abdominal muscle layers will be identified, and the transverses abdominis plane will be located between the internal oblique and the transverse abdominis muscle. The TAP will be approached through in-plane technique using a 23-gauge Quincke spinal needle attached to a 20 ml syringe of 0.25% bupivacaine will be injected and the drug spread in the plane will be observed. The same procedure will be repeated on the other side of the abdomen.

In ILIH group, the probe will be placed medial to the lateral one-third of the line joining the umbilicus and the anterior superior iliac spine (ASIS), with part of the probe sitting on the ASIS. The ASIS, iliacus muscle, internal oblique, transverses abdominis, and the ILIH nerves between them will be identified. After appreciating the sonoanatomy, the ILIH nerve will be approached with the 23-gauge Quincke spinal needle through in-plane technique and 10 ml of 0.25% bupivacaine will be injected all around and the drug spread will be appreciated. The same procedure will be repeated on the other side.

For the QLB, the transducer will be placed at the level of the anterosuperior iliac spine and will move cranially until the 3 abdominal wall muscles will be clearly identified. The external oblique muscle will be followed posterolaterally until its posterior border was visualized (hook sign), leaving underneath the internal oblique muscle, like a roof over the quadratus lumborum muscle. The probe will be tilted down to identify a bright hyperechoic line that corresponded with the middle layer of he thoracolumbar fascia. The needle (21 gauge) will be inserted in plane from anterolateral to posteromedial. The optimal point of injection for the QL block will be determined over the lumbar interfacial triangle using hydrodissection.

At the end of the procedure, patients will be shifted to the postanesthesia recovery room and later to the postoperative ward after establishing the block.

The sensory assessment following the TAP, ILIH, and QLB block will be done after confirming the spinal regression below the level of L2 dermatome. The block will be considered "Successful" when the patient will not be able to perceive the cold sensation at L1 dermatome (inguinal region) on both sides. The block will be considered "Partial" when patient perceives cold sensation on any one of the side.

The block will be considered "Failure" when the patient perceives cold sensation on both sides at L1 dermatome. Patients suffering partial and failed block will be excluded from the study for further analysis but will receive standard postoperative analgesics as any other patients. In the postoperative ward, whenever, the patient complained of pain, nurse in-charge will note the numerical rating scale (NRS) score, and will administered a single dose of injection diclofenac sodium of 50 mg as slow intravenous infusion over a period of 15 min and will note the time as time of first analgesia. Subsequently, whenever patient complain of pain, injection tramadol 50 mg will be given intravenously for the remaining 24 h.

A blinded observer who will not be aware of the group allocation will visit the patient at 2, 4, 6, 10, 12, and 24 h postoperative intervals and analyz the study parameters and record in the common standard data nalogue scale for pain (ranging from 0 to 10 with 0 no pain, 10 being severe pain, and the patients will be asked to mark the pain score on the scale) during rest as well as on movement (turning lateral to any one side). Duration of analgesia will be taken as time interval between the block time and the time of first analgesia.

The 24 h requirement of rescue analgesics injection diclofenac sodium and injection tramadol and complications such as nausea, vomiting, transient femoral nerve palsy, any signs, and symptoms of bowel perforation will be noted.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1 and 2
* Aged between 18 and 45 years
* Scheduled for emergency or elective lower segment cesarean section

Exclusion Criteria:

* Pregnant women who will refuse to participate.
* Known allergy to local anesthetic.
* Infection at the block site.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
The quality of analgesia | 2 hours postoperatively
  The quality of analgesia was assessed by NRS (unidimensional 11-point pain scale ranging from 0 to 10 with 0 no pain, 10 being severe pain, and the patients will be asked to mark the pain score on the scale)
The quality of analgesia | 4 hours postoperatively
  The quality of analgesia was assessed by NRS (unidimensional 11-point pain scale ranging from 0 to 10 with 0 no pain, 10 being severe pain, and the patients will be asked to mark the pain score on the scale)
The quality of analgesia | 6 hours postoperatively
  The quality of analgesia was assessed by NRS (unidimensional 11-point pain scale ranging from 0 to 10 with 0 no pain, 10 being severe pain, and the patients will be asked to mark the pain score on the scale)
The quality of analgesia | 10 hours postoperatively
  The quality of analgesia was assessed by NRS (unidimensional 11-point pain scale ranging from 0 to 10 with 0 no pain, 10 being severe pain, and the patients will be asked to mark the pain score on the scale)
The quality of analgesia | 12 hours postoperatively
  The quality of analgesia was assessed by NRS (unidimensional 11-point pain scale ranging from 0 to 10 with 0 no pain, 10 being severe pain, and the patients will be asked to mark the pain score on the scale)
The quality of analgesia | 24 hours postoperatively
  The quality of analgesia was assessed by NRS (unidimensional 11-point pain scale ranging from 0 to 10 with 0 no pain, 10 being severe pain, and the patients will be asked to mark the pain score on the scale)